CLINICAL TRIAL: NCT04956198
Title: Drug Sensitivity Testing and Mutation Profiling in Childhood Sarcomas
Brief Title: Drug Sensitivity and Mutation Profiling
Status: Completed | Type: Observational
Sponsor: Florida International University (Other)
Collaborators: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); Cornelia T. Bailey Foundation (Unknown)
Responsible Party: Principal Investigator, Diana Azzam, PhD, Assistant Professor, Florida International University
Other Study IDs: 1294510
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Ewing Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Wilms Tumor; Sarcoma, Spindle Cell; Sarcoma Rhabdoid; Childhood Sarcoma of Soft Tissue
Keywords: ex vivo drug sensitivity assay; genomic profiling
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Wilms Tumor; Sarcoma; Rhabdoid Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Perform molecular and functional drug testing on blood, biopsy, bone marrow, and tumor samples at relapse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with newly diagnosed as well as relapsed/refractory sarcomas.: The investigators intend to enroll newly diagnosed or refractory/relapsed pediatric patients with all types of sarcomas where tumor tissue would be available for ex vivo drug screening and genomic profiling. This observational study will assess how ex vivo drug testing and mutation profiling may predict clinical outcomes (response, survival, or relapse). The treating physician will decide which of the standard treatment options is appropriate independent of the DST results. The results of DST will not be available to the treating physician at the time of decision on the treatment regimen. DST will include all drugs from the standard treatment regimens available for all types of sarcomas

SUMMARY:
This study is a prospective, non-randomized observational study. Freshly isolated tumor cells will be tested for chemosensitivity to the standard of care drugs as single agents and in combinations using state-of-the-art viability assay designed for ex-vivo high-throughput drug sensitivity testing (DST). In addition, the genetic profile of the tumor will be obtained from the medical records and correlated with drug response.

DETAILED DESCRIPTION:
The excised tumors or a biopsy will be interrogated for sensitivity or resistance to FDA-approved and/or available investigational agents. In addition, normal samples (blood or buccal swab) will be collected for genetic analysis of germline mutations and cancer predisposition markers. The timeframe between the sample acquisition and ex vivo DST results return will be approximately 5-10 working days. All drugs tested in the DST assay will be assigned a hybrid score reflecting the tumor's sensitivity and drug toxicity.

This is an observational study and not a treatment protocol. It will assess how ex vivo drug testing and mutation profiling may predict clinical outcomes (response, survival, or relapse). The treating physician will decide which of the standard treatment options is appropriate independent of the DST results. The results of DST will not be available to the treating physician at the time of decision on the treatment regimen. DST will include all drugs from the standard treatment regimens available for all types of sarcomas

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or younger at the time of enrollment on this study of any gender, race, or ethnicity.
* Subjects with suspected or confirmed diagnosis of all types of sarcomas.
* Subjects who are scheduled for or have recently had biopsy or tumor excised (solid tumors) or bone marrow aspirate (blood cancers).
* Subjects are willing to have a blood draw or buccal swab done for the purposes of genetic testing.
* Subjects or their parents or legal guardians willing to sign informed consent.
* Subjects aged 7 to 17 willing to sign assent.

Exclusion Criteria:

* Subjects who do not have malignant tissue available and accessible.
* The amount of excised malignant tissue is not sufficient for ex vivo drug testing and/or genetic profiling.
* Patients with other types of tumors and tumors that have a high (>90%) cure rate with safe standard therapy.

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with newly diagnosed as well as relapsed/refractory sarcomas.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To correlate results of drug sensitivity and mutation profiles with clinical outcomes in response to therapy. | Up to 4 years
  Response to therapy (RTT): an event of achieving "partial response" or "complete response" during the study period, based on the best response of the corresponding enrolled patient.
To correlate results of drug sensitivity and mutation profiles with clinical outcomes in progression-free survival. | Up to 4 years
  Progression-free survival (PFS): a composite end point defined as the censored event time from enrollment to either disease relapse or mortality. This will be evaluated retrospectively at the end of the study. The investigators will use the two-sample long-rank test to assess the hazard ratio of PFS events between the two groups classified as drug sensitive and insensitive by the DST.The study will enroll 15 patients and it is assumed 50% of these subjects will be classified as drug sensitive based on the DST at the threshold value of 10.

SECONDARY OUTCOMES:
To assess the predictive value of personalized approach in predicting RTT. | Up to 4 years
  Classification accuracy of DST for predicting the RTT
To assess the predictive value of personalized approach in predicting PFS. | Up to 4 years
  Classification accuracy of DST for predicting the PFS
  The DTS test results will be treated as the continuous classifier, and the binary RTT status for each subject along with the binary PFS status by the end of the study will be used as the binary reference status (with and without RTT/PFS endpoint). The area under the curve (AUC) of the resulting ROC curve will be used a metric for the overall classification accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Diana Azzam, PhD, Principal Investigator — Florida International University; Daria Salyakina, PhD, Principal Investigator — Nicklaus Children's Hospital; Maggie Fader, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States